CLINICAL TRIAL: NCT05965739
Title: RECOVER-NEURO: A Platform Protocol for Evaluation of Interventions for Cognitive Dysfunction in Post-Acute Sequelae of SARS-CoV-2 Infection (PASC)
Brief Title: RECOVER-NEURO: Platform Protocol, Appendix_A to Measure the Effects of BrainHQ, PASC CoRE and tDCS Interventions on Long COVID Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00112477_A; OTA-21-015G (Other Grant/Funding Number: NIH grant to RTI; RTI subcontracting with DCRI); 1OT2HL156812-01 (NIH)
Record Dates: First submitted 2023-07-25; First posted 2023-07-28 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-02

CONDITIONS: Long COVID; Long Covid19; Long Covid-19
Keywords: PASC; Cognitive
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: To achieve blinding and an equitable randomization probability, a two-step randomization process will be used. The study will employ a simple (unstratified) randomization scheme.
  At the first stage, each participant will be assigned with equal probability to one of the intervention appendices for which the participant is eligible, after applying any intervention-specific safety exclusions. At the second stage, each participant will be assigned according to the specific appendix's randomization procedure. Participants will have an equal chance of being randomized into any of the intervention groups.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants assigned to control will be considered part of pooled analyses if the intervention was active at the time of their enrollment and the participants were eligible to receive that intervention. This will result in approximately a 1:1 allocation ratio for any intervention to pooled control.
  Sites will be informed to which intervention appendix participants are randomized, but, when applicable, not whether the participants are allocated to the active intervention arm or control arm within that appendix. The participants and investigators will be blinded throughout the study, when possible.
  If open intervention appendices do not have the ability to pool controls but have independent controls, at the second stage participants will be randomized in a 1:1 ratio to intervention vs control inside the specific intervention appendix the participants were randomized to at the first stage of the randomization procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- BrainHQ Active Comparator (Active Comparator): 5 sessions/week at 30 min/session
  Interventions: Other: BrainHQ/Active Comparator Activity
- BrainHQ (Experimental): 5 sessions/week at 30 min/session
  Interventions: Other: BrainHQ
- BrainHQ + PASC CoRE (Experimental): BrainHQ plus 9 group sessions at 1.5 hr/session and 3 individual sessions at 1 hr/session
  Interventions: Other: BrainHQ; Other: PASC CoRE
- Brain HQ + tDCS-active (Experimental): 2.0 mA stimulation delivered for 30 min during each BrainHQ session
  Interventions: Other: BrainHQ; Device: tDCS-active
- Brain HQ + tDCS-sham (Placebo Comparator): Inactive stimulation delivered for 30 min during each BrainHQ session
  Interventions: Other: BrainHQ; Device: tDCS-sham

INTERVENTIONS:
Other: BrainHQ/Active Comparator Activity — BrainHQ platform provides a set of cognitive activities, like puzzles and games, that are cognitively stimulating and actively engage participants but do not continuously and adaptively challenge them. These activities are designed to be a face-valid, active comparison approach to cognitive therapy, thus participants are blinded, attention time is matched, and overall user experience is identical to the active arms.
  Arms: BrainHQ Active Comparator
Other: BrainHQ — BrainHQ is an online cognitive training program, and has been used to improve cognitive function among persons with cognitive impairment based on principles of neuroplasticity.
  Arms: Brain HQ + tDCS-active; Brain HQ + tDCS-sham; BrainHQ; BrainHQ + PASC CoRE
Other: PASC CoRE — PASC CoRE is a manualized, adaptable cognitive rehabilitation intervention adapted from Goal Management Training and other evidence based programs that improve attention and executive functions, among other cognitive domains.
  Arms: BrainHQ + PASC CoRE
Device: tDCS-active — Transcranial direct current stimulation (tDCS) will use a device specifically for home-based use. This device delivers a weak electrical current of 2.0 mA passed through two electrodes placed on the scalp to target the dorsolateral prefrontal cortex region of the brain. The electrodes are single-use for each session and can be attached to a headset by snapping into place.
  The device has a user-friendly interface and a large-button keypad, making it is easy to use at home.
  Arms: Brain HQ + tDCS-active
Device: tDCS-sham — tDCS devices used in the sham arm will be pre-programmed to deliver the same ramp up/down at the beginning/end of the 30-minute period as the active arm, except with no current otherwise delivered during the session.
  Arms: Brain HQ + tDCS-sham

SUMMARY:
This platform protocol is designed to be flexible so that it is suitable for a wide range of settings within health care systems, for remote settings, and in community settings where it can be integrated into COVID-19 programs and subsequent treatment plans.

This protocol is a prospective, multi-center, multi-arm, randomized, controlled platform trial evaluating potential interventions for PASC-mediated cognitive dysfunction. The hypothesis is that PASC-associated dysfunction in cognitive domains, such as executive function and attention, may be improved by interventions that selectively focus on enhancing those domains.

This design seeks to evaluate each intervention relative to the Active Comparator. The BrainHQ (alone) arm is important because the intervention is commercially available, accessible, relatively inexpensive, and does not require trained personnel to administer. BrainHQ has been also been proven effective in other studies of cognitive dysfunction such as studies in aging, mild cognitive impairment, traumatic brain injury, among others. The BrainHQ + PASC CoRE arm and the BrainHQ + tDCS arms are suspected to provide cognitive improvements beyond BrainHQ alone through different mechanisms. Both PASC CoRE and tDCS have extensive prior use and have demonstrated utility in improving aspects of cognitive function in other clinical settings..

DETAILED DESCRIPTION:
Participants will be randomized to one of the intervention appendices that are actively enrolling at the time of randomization. Intervention appendices may be added or removed according to adaptive design and/or emerging evidence. Various interventions will be studied.

Participants will be randomized equally across the five arms:

1. Active Comparator (video games)
2. BrainHQ
3. BrainHQ + PASC CoRE
4. BrainHQ + tDCS-active
5. BrainHQ + tDCS-sham

ELIGIBILITY:
Inclusion Criteria:

1. See NCT05965752 for RECOVER-NEURO: Platform Protocol level inclusion criteria which applies to this appendix

Exclusion Criteria:

1. See NCT05965752 for RECOVER-NEURO: Platform Protocol level exclusion criteria which applies to this appendix

Additional Appendix (Sub-study) Level Exclusion Criteria:

1. Presence of metal objects in the head or neck
2. Skin disorders or skin-sensitive areas near tDCS stimulation locations that would interfere with electrode placement or increase the risk of stimulation-induced damage, at the investigator's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Change in Everyday Cognition 2 (ECog2) | Baseline to End of Intervention (EOI) (Day 70)
  Everyday Cognition 2 (ECog2) is a self-report, 41-item questionnaire used to measure the participant's simple reaction time; respond when X happens and Choice reaction time; respond only if X happens.

SECONDARY OUTCOMES:
Change in PROMIS-cognitive function - short form 8a (PROMIS-Cog) total score | Baseline, EOI (Day 70), End of Study (EOS) (Day 160)
  The PROMIS-Cog is the PROMIS short form for the cognitive function domain and is a self-report, 8-item questionnaire targeting cognitive function in the past seven days.
Change on an objective neurocognitive battery scores | Baseline, EOI (Day 70), EOS (Day 160)
Change in Everyday Cognition 2 (ECog2) | Baseline, EOS (Day 160)
  Everyday Cognition 2 (ECog2) is a self-report, 41-item questionnaire used to measure the participant's simple reaction time; respond when X happens and Choice reaction time; respond only if X happens.
Characterize the intervention's safety as measured by the proportion of Serious Adverse Events, Unanticipated Adverse device Effects, and/or Events of Special Interest [Proportion of SAEs, UADEs, and/or ESIs.] | Baseline to EOS (Day 160)

CONTACTS AND LOCATIONS:
Overall Officials: Kanecia Zimmerman, MD PhD, Study Chair — Duke University; Daniel Laskowitz, MD MHS, Study Chair — Duke University
Locations (1):
- All sites listed under NCT05965752, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The investigators will share the summary of results on the study website: https://recovercovid.org/

REFERENCES:
- [Derived] Knopman DS, Koltai D, Laskowitz DT, Becker J, Charvet L, Wisnivesky J, Federman A, Silverstein A, Lokhnygina Y, Pilloni G, Haddad M, Mahncke H, Van Vleet T, Huang R, Cox W, Terry D, Karwowski J, McCray N, Lin JJ, McComsey GA, Singh U, Geng LN, Chu HY, Reece R, Moy J, Arvanitakis Z, Parthasarathy S, Patterson TF, Gupta A, Ostrosky-Zeichner L, Parsonnet J, Kiriakopoulos ET, Fong TG, Mullington J, Jolley S, Shah NS, Morimoto SS, Lee-Iannotti JK, Killgore WDS, Dwyer B, Stringer W, Isache C, Frontera JA, Krishnan JA, O'Steen A, James M, Harper BL, Zimmerman KO; RECOVER-NEURO Clinical Trial Group. Evaluation of Interventions for Cognitive Symptoms in Long COVID: A Randomized Clinical Trial. JAMA Neurol. 2026 Jan 1;83(1):49-59. doi: 10.1001/jamaneurol.2025.4415. PMID 41212544
- [Derived] Knopman DS, Laskowitz DT, Koltai DC, Charvet LE, Becker JH, Federman AD, Wisnivesky J, Mahncke H, Van Vleet TM, Bateman L, Kim DY, O'Steen A, James M, Silverstein A, Lokhnygina Y, Rich J, Feger BJ, Zimmerman KO. RECOVER-NEURO: study protocol for a multi-center, multi-arm, phase 2, randomized, active comparator trial evaluating three interventions for cognitive dysfunction in post-acute sequelae of SARS-CoV-2 infection (PASC). Trials. 2024 May 17;25(1):326. doi: 10.1186/s13063-024-08156-z. PMID 38755688
- See also: Related Info — http://recovercovid.org/

DOCUMENTS (1):
  • Informed Consent Form (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/39/NCT05965739/ICF_000.pdf